CLINICAL TRIAL: NCT00549276
Title: Randomized Comparison of Curved Cutter Stapler and Linear Stapler
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Other Study IDs: Samsung Medical Center
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2006-05

CONDITIONS: Rectal Neoplasm; Surgical Stapler
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to compare the safty and technical accessibility of linear stapler and curved cutter stapler during mid to low rectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of rectum.
* Preoperative stage I-III
* Patient who is expected to undergo low anterior resection at Samsung Medical Center.
* Age > 19 years old

Exclusion Criteria:

* Patient with complicated rectal cancers(obstruction, perforation, abscess)
* Patient who needs to undergo emergency operation.
* Patient who can not undergo general anesthesia.
* Patient who does not agree with the informed consent or does not have the ability to understand content of the trial .

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients were randomly assigned to either linear staplers or the CCS during low anterior resection for mid to low rectal cancers
Sampling Method: Probability Sample
Dates: Start 2006-05; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Suk Lee, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center Sungkyunkwan University School of Medicine,, Seoul, South Korea